CLINICAL TRIAL: NCT02404402
Title: Noninvasive LED Treatment to Improve Cognition and Promote Recovery in Blast TBI
Brief Title: LED Treatment to Improve Cognition and Promote Recovery in TBI
Acronym: LED-TBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N1773-P
Record Dates: First submitted 2015-02-25; First posted 2015-03-31 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorder
Keywords: Traumatic Brain Injury; Light Emitting Diodes; Cognition; Neuromodulation; PTSD; Neurorehabilitation; Veterans; Sleep
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active LED (Experimental): Active LED Treatment
  Interventions: Other: LED
- Sham LED (Sham Comparator): Inactive (sham) LED Treatment
  Interventions: Other: sham LED

INTERVENTIONS:
Other: LED — Low Level Light Therapy
  Arms: Active LED
Other: sham LED — Inactive (sham) LED treatment
  Arms: Sham LED

SUMMARY:
This study investigates the efficacy of a novel neuromodulation treatment, light emitting diodes (LED), on cognition, neuropsychiatric status and quality of life in individuals with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
The most common traumatic brain injury (TBI)-associated problems are cognitive deficits and neuropsychiatric problems, such as sleep disturbance and PTSD. This study evaluates a novel neuromodulation intervention, light emitting diodes (LED), for treatment of patients with TBI. LED is a noninvasive, non-thermal, painless treatment, which does not involve any needles or any form of surgery. LED treatment improves cellular activity of the brain tissue that has been damaged by TBI. Half of the study participants will receive active LED treatment, and a control group will receive sham LED. This study takes place in Boston, Massachusetts: at the VA Boston Healthcare System.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* OEF/OIF active-duty personnel or Veterans with history of TBI or blast-exposure
* Meets criteria for mild TBI
* LOC of 30 min or less
* Age: 21-55
* Primary language is English

Exclusion Criteria:

* Evidence of penetrating head injury
* History of previous neurological diagnosis
* History of previous psychotic disorder prior to TBI
* Hearing or vision impairment

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functioning_Attention/Executive | Eight Weeks
  Stroop Test ("Color-Word" test; Delis, Kaplan & Kramer, 2001)
Cognitive Functioning_Learning/Memory | Eight weeks
  California Verbal Learning Test-II (CVLT-II; Delis, Kramer, Kaplan, & Ober, 2000)

SECONDARY OUTCOMES:
Neuropsychiatric Status/Mood | Eight weeks
  Beck Depression inventory (BDI; Beck, 2006)
Neuropsychiatric status/PTSD | Eight weeks
  PTSD Checklist - Military Version (PCL-M)
Neuropsychiatric status/Sleep | Eight weeks
  Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Bogdanova, PhD PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No